CLINICAL TRIAL: NCT06049459
Title: Novel Amblyopia Treatment With Dichoptic, Disparity-guided, Hand-Eye Coordination Enhanced, Serious, Virtual Reality Games
Brief Title: Novel Amblyopia Treatment With Virtual Reality Games
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marjean Kulp (Other)
Collaborators: Beta Sigma Kappa - College of Optometrists in Vision Development (Unknown); VividVision (Unknown)
Responsible Party: Sponsor-Investigator, Marjean Kulp, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023H0013
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: This is a within-subject study, and all participants complete both study conditions. Each participant completes 16 weeks of optical correction alone (if needed) followed by 16 weeks of Therapeutic (Dichoptic) Virtual Reality Games plus continued optical correction. Each subject serves as their own control.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be masked to past performance and adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Optical Correction alone (Active Comparator): Optical correction alone (16 weeks) (Each participant will complete both study conditions.)
  Interventions: Device: Optical Correction
- Therapeutic (Dichoptic) Virtual Reality Games plus Continued Optical Correction (Experimental): Therapeutic (Dichoptic) Virtual Reality Games plus continued optical correction (16 weeks) (Each participant will complete both study conditions.)
  Interventions: Device: Optical Correction; Device: Therapeutic Dichoptic Virtual Reality Games

INTERVENTIONS:
Device: Optical Correction — Optical correction (if needed)
Device: Therapeutic Dichoptic Virtual Reality Games — Virtual Reality Game play for amblyopia treatment
  Arms: Therapeutic (Dichoptic) Virtual Reality Games plus Continued Optical Correction

SUMMARY:
The goal of this study is to compare the change in amblyopic eye acuity between treatment periods in children with amblyopia, aged 5-17 years. The main question it aims to answer is:

Is a 16-week course of amblyopia treatment using Vivid Vision Therapeutic (Dichoptic) Virtual Reality Games for approx. 25 min/day, 6 days/week more effective for improvement in amblyopic-eye VA, binocularity (stereoacuity, suppression, alignment), contrast sensitivity, attention, oculomotor function, visual-motor integration, and quality of life than 16 weeks of continued glasses alone?

Participants will each serve as their own control and complete:

Treatment period 1: Continued optical correction (glasses) alone for 16 weeks; Treatment period 2: Vivid Vision Therapeutic (Dichoptic) Virtual Reality Games for 16 weeks (approx. 25min/day, 6 days/week) plus continued optical correction

ELIGIBILITY:
Inclusion Criteria:

Patients ages 5 to 17 years of age

* Moderate to severe unilateral amblyopia (logMAR best corrected visual acuity 0.3 to 1.3) associated with anisometropia and/or strabismus of ≤5pd
* Age normal VA in the nonamblyopic eye
* Spectacle correction (if required) worn for at least 16 weeks, or until stability of VA is demonstrated (<0.1 logMAR change by the same testing method measured on 2 exams at least 8 weeks apart)
* Interocular difference of ≥ 3 lines
* No amblyopia treatment in the past 2 weeks
* An interpupillary distance of 52-72 mm (inclusive)

Exclusion Criteria:

* Myopia greater than -6.00 diopters (D) spherical equivalent in either eye.
* Previous intraocular or refractive surgery.
* Previous dichoptic treatment > 2 weeks in duration
* Ocular co-morbidity that may reduce visual acuity determined by an ocular examination performed within the past 7 months (Note: nystagmus per se does not exclude the participant if the above visual acuity criteria are met).
* Diplopia more than once per week over the last week prior to enrollment by parental report.
* Down syndrome or cerebral palsy.
* Light-induced seizures
* Known simulator sickness
* Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities are not excluded.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Mean Change in Amblyopic Eye Visual Acuity | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Optical correction worn for testing using Amblyopia Treatment Study (ATS) protocol; HOTV for ages 5-6 years; E-ETDRS for ages 7 years and older

SECONDARY OUTCOMES:
Difference in Change in Stereoacuity/Binocularity | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Optical correction worn for testing. Stereoacuity scores (seconds of arc) calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) tests. Lower scores indicate better stereoacuity. Nil (4000) defined as an incorrect response (or lack of an attempt) on the butterfly without a correct response on 800 seconds of arc level of Randot Preschool stereoacuity test. Stereoacuity scores will be ordered and assigned a rank score. Change in stereoacuity will be calculated as the difference in change in ranked score.
Difference in Mean Change in Amblyopic-Eye Contrast Sensitivity | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Optical correction worn for testing. Spot Checks;Contrast sensitivity scores range from unable (<0.90), and then from 0.90 to 2.05 (by 0.05 log contrast sensitivity units).
Difference in Mean Change in Attention | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Optical correction worn for testing. The Children's Color Trails Test (CCTT) is a neuropsychological standardized test that measures attention, divided attention, and speed of mental processing.
Difference in Mean Change in reading eye movements | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Optical correction worn for testing with Readalyzer eye tracker.
Difference in Mean Change in visual-motor integration | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Optical correction worn for testing. Beery Visual-Motor Integration; standard scores with mean of 100, standard deviation of 15
Difference in Mean Change in Pediatric Eye Questionnaire (PedEyeQ) | Baseline to 16 weeks versus 16 weeks to 32 weeks
  Pediatric Eye Questionnaire (PedEyeQ) domain score; scores for questionnaire items will be obtained from published look-up tables available at www.pedig.net; scaled to score from 0 to 100 (worst to best)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No